CLINICAL TRIAL: NCT02362763
Title: The Use of Acupuncture for the Treatment of Vulvar Vestibulitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, hamaniHMO, Dr. Yaron Hamani, Hadassah Medical Organization
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VESTIB-HMO-CTIL
Record Dates: First submitted 2015-01-28; First posted 2015-02-13 (Estimated); Last update posted 2015-02-13 (Estimated); Status verified 2015-02

CONDITIONS: Vestibulodynia
MeSH Terms: conditions — Vulvodynia | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Study group (Experimental): Subjects received five acupuncture sessions designed to treat pain in the vulvar area
  Interventions: Procedure: Acupuncture
- Controls (Active Comparator): Controls received five acupuncture sessions designed for sedation
  Interventions: Procedure: Acupuncture

INTERVENTIONS:
Procedure: Acupuncture — Patients randomized to the study group received five sessions of acupuncture in a series of points in the lower abdomen, lower back, hands, and feet. This combination of acupoints is believed to impact on the genital area, raise the pain threshold, and counteract inflammation. Control group patients received five sessions of acupuncture at acupoints that are believed to have no influence on the genital area, but are believed to have a general sedative effect.

SUMMARY:
Randomized controlled trial designed to determine whether acupuncture is an effective treatment for vestibulitis.

DETAILED DESCRIPTION:
Patients were randomized to five acupuncture sessions designed to treat pain in the vulvar area (study group), or five acupuncture sessions designed for tranquility (controls). Participants and evaluating gynecologists were blinded to randomization. Participants were examined clinically before treatment and one month after completion of assigned treatment; at both visits they completed the Female Sexual Function Index (FSFI) questionnaire.

FSFI scores for pain during intercourse and total score were used to evaluate change. The examining gynecologist evaluated the degree of sensitivity to touch and the degree of local erythema. Response to treatment was evaluated for each group before and after treatment, and for study group compared to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of vestibulodynia

Exclusion Criteria:

* Pregnancy
* Patient who received other treatment for vestibulodynia in the month preceding.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2006-06; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Female Sexual Function Index (FSFI) questionnaire | 1 month after completion of the assigned treatment

SECONDARY OUTCOMES:
Clinical examination | 1 month after completion of the assigned treatment
  Visual presence or absence of vestibular erythema

CONTACTS AND LOCATIONS:
Overall Officials: Yaron Hamani, MD, Principal Investigator — Hadassah Medical Organization